CLINICAL TRIAL: NCT03789162
Title: Blood and Stool Sample Collection in Subjects With a Diagnosis of Colorectal Cancer or Colorectal Lesion: Act Fast
Status: Completed | Type: Observational
Sponsor: Exact Sciences Corporation (Industry)
Responsible Party: Sponsor
Other Study IDs: 2018-07
Record Dates: First submitted 2018-12-18; First posted 2018-12-28 (Actual); Last update posted 2025-06-29 (Actual); Status verified 2025-06

CONDITIONS: Colorectal Cancer
Keywords: Blood Draw; Sample Collection; Stool DNA
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Specimens collected under this protocol may be stored indefinitely for future research in addition to and separate from the study and use of specimens and data described in the rest of this protocol. Specimens are de-identified of all protected health information and clinical study data will only be associated by a subject identification number. Specimens de-accessioned from the biorepository will be destroyed under standard biohazardous material protocol and record of the removal and destruction will be maintained for 7 years by the Sponsor. Specimens and/or data collected during this study may be used by the Sponsor and its affiliates and may also be shared with and used by other outside individuals and organizations.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Confirmed CRC with Residual Lesion: A diagnosis of CRC confirmed with a tissue biopsy or a colorectal lesion at least 1 cm in size suspicious for adenoma (including sessile serrated adenoma) or CRC on a pre-enrollment colonoscopy.

SUMMARY:
The primary objective of this study is to collect de-identified, clinically-characterized stool and whole blood specimens for use in developing and evaluating the performance of new biomarker assays for the detection of colorectal cancer (CRC).

DETAILED DESCRIPTION:
Participants will be 40 years of age or older, with a diagnosis of CRC, at any stage, confirmed with a tissue biopsy or a colorectal lesion at least 1 cm in size suspicious for adenoma (including sessile serrated adenoma) or CRC on a pre-enrollment colonoscopy, sigmoidoscopy, or computed tomography (CT) colonography. Approximately 1500 participants will be enrolled.

ELIGIBILITY:
Inclusion Criteria:

1. Participant is 40 years of age or older.
2. Participant has a diagnosis of CRC, at any stage, confirmed with a tissue biopsy or a colorectal lesion at least 1 cm in size suspicious for adenoma (including sessile serrated adenoma) or CRC on a pre-enrollment colonoscopy, sigmoidoscopy, or CT colonography.
3. Postcolonoscopy, the residual lesion in the colon must be at least 1 cm in size as to require additional surgical excision or complex colonoscopic polypectomy.
4. Participant understands the study procedures and is able to provide informed consent to take part in the study and authorization for release of relevant protected health information to the study Investigator.

Exclusion Criteria:

1. Any previous cancer diagnosis (with the exceptions of basal cell or squamous cell skin cancers) and/or cancer related treatment (e.g., chemotherapy, immunotherapy, radiation, and/or surgery) within the past 5 years.
2. Less than 7 days between colonoscopy and blood and/or stool specimen collection.
3. IV contrast (e.g., CT or MRI) within 1 day [or 24 hours] before blood and/or stool collection.
4. Participant has any condition that in the opinion of the Investigator should preclude taking part in the study.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Approximately 1500 subjects will be enrolled. Participants will be 40 years of age or older, with a diagnosis of CRC, at any stage, confirmed with a tissue biopsy or a colorectal lesion at least 1 cm in size suspicious for adenoma (including sessile serrated adenoma) or CRC on a pre-enrollment colonoscopy, sigmoidoscopy, or computed tomography (CT) colonography.
Sampling Method: Non-Probability Sample
Enrollment: 850 (Actual)
Dates: Start 2018-12-20 (Actual); Primary Completion 2025-03-31 (Actual); Study Completion 2025-05-29 (Actual)

PRIMARY OUTCOMES:
Stool-based biomarkers associated with genetic and epigenetic alterations | Stool sample will be collected at least 7 days after the subject's pre-enrollment colonoscopy, but prior to initiation of bowel preparation for any follow-up procedure
  The outcomes are co-primary. Biomarkers under evaluation include differential methylation of nucleic acids and altered expression of proteins in stool from subjects with confirmed colorectal cancer at the pre-intervention stage.
Blood-based biomarkers associated with genetic and epigenetic alterations | Point in time blood collection (1 day) at enrollment
  The outcomes are co-primary. Biomarkers under evaluation include differential methylation of nucleic acids and altered expression of proteins in blood from subjects with confirmed colorectal cancer at the pre-intervention stage.

CONTACTS AND LOCATIONS:
Locations (45):
- United States (44):
  - Mayo Clinic - Arizona, Phoenix, Arizona
  - Alliance Research Institute, Canoga Park, California
  - GW Research Inc, Chula Vista, California
  - Tilda Research, Laguna Hills, California
  - Clinical Trials Network, San Diego, California
  - Gastroenterology Associates of Fairfield County, P.C., Fairfield, Connecticut
  - Connecticut Clinical Research Institute, Hartford, Connecticut
  - Yale University, New Haven, Connecticut
  - Guardian Angel Research Center, Tampa, Florida
  - Rush University Medical Center, Chicago, Illinois
  - DM Clinical Research/Southwest Gastroenterology, Oak Lawn, Illinois
  - Southern Illinois University School of Medicine, Springfield, Illinois
  - Carle Foundation Hospital dba Carle Cancer Center, Urbana, Illinois
  - Deaconess Clinic, Inc., Evansville, Indiana
  - Digestive Research Alliance of Michiana, LLC, South Bend, Indiana
  - MZS Research, LLC, Metairie, Louisiana
  - Delta Research Partners, Monroe, Louisiana
  - Louisiana Research Center, LLC, Shreveport, Louisiana
  - Clinical Trials of America, LLC, West Monroe, Louisiana
  - Capitol Research, Rockville, Maryland
  - HealthPartners Institute, Saint Louis Park, Minnesota
  - Park Nicollet Oncology Research, Saint Louis Park, Minnesota
  - Virtua Health Inc, Marlton, New Jersey
  - University Health Service Hospitals, Inc., Binghamton, New York
  - Icahn School of Medicine at Mount Sinai Beth Israel, New York, New York
  - Digestive Health Partners, PA, Asheville, North Carolina
  - Charlotte Gastroenterology & Hepatology, PLLC, Charlotte, North Carolina
  - Trial Management Associates, LLC, Wilmington, North Carolina
  - Clinical Trials Network, Beachwood, Ohio
  - Clinical Trials Network, Mentor, Ohio
  - Susquehanna Research Group, Camp Hill, Pennsylvania
  - Frontier Clinical Research, LLC, Uniontown, Pennsylvania
  - Spartanburg Regional Health Services District, Inc, Spartanburg, South Carolina
  - Digestive Health Research, LLC, Hermitage, Tennessee
  - The Jackson Clinic Professional Association, Jackson, Tennessee
  - Advanced Gastroenterology, Union City, Tennessee
  - Northside Gastroenterology Associates PA, Cypress, Texas
  - Digestive Health, Houston, Texas
  - The University of Texas Health Science Center at Houston, Houston, Texas
  - Texarkana Clinical Research, Texarkana, Texas
  - Blue Ridge Medical Research, Lynchburg, Virginia
  - Virginia Gastroenterology Institute, Suffolk, Virginia
  - MultiCare Institute for Research & Innovation - Tacoma, Tacoma, Washington
  - HSHS St. Vincent Hospital Regional Cancer Center, Green Bay, Wisconsin
- University of Clagary, Forzani & MacPhail Colon Cancer Screening Centre, Calgary, Alberta, Canada

IPD SHARING:
Plan to Share IPD: No